CLINICAL TRIAL: NCT06218329
Title: TIMECARD (TaIwan Network of Post-arrest ManagEment for CARDiac Arrest) II Registry
Brief Title: TIMECARD(TaIwan Network of Post-arrest ManagEment for CARDiac Arrest)IIRegistry
Acronym: TIMECARDII
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Clinical Trial Center (Other)
Responsible Party: Sponsor-Investigator, National Taiwan University Clinical Trial Center, National Taiwan University Hospital, National Taiwan University Hospital
Organization: National Taiwan University Hospital (Other)
Other Study IDs: 202201091RINB
Record Dates: First submitted 2023-10-17; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2023-10

CONDITIONS: Cardiology, Critical Care Medicine, Emergency Medical Service
Keywords: Prognosis, post-cardiac arrest syndrome, Sudden Cardiac Arrest, registry database, predictive model
MeSH Terms: conditions — Post-Cardiac Arrest Syndrome; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to collect the post-cardiac arrest patients with ICU admission.

DETAILED DESCRIPTION:
The purpose of this study is to establish protocolized and standard post-arrest care as well as constitute a multicenter registry of post-arrest survivors, and thus to develop the Taiwan predictive model of cardiac arrest survivors. The registry system may help evaluate the severity of disease illness and improve the post-arrest care.

ELIGIBILITY:
Inclusion Criteria:

* non-traumatic cardiac arrest patients
* Admitted to the ICU

Exclusion Criteria:

* Below 18 year old
* Pregnant
* Terminal illness or not receiving medical treatment
* When emergency ICU crowded can not provide Critical Care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients with who arrived at the emergency department with non-traumatic and admitted to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of cases | 2024/12/31

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Emergency Medicine, National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No